CLINICAL TRIAL: NCT06992635
Title: Effect of Smart Phone Reflective Light Film on Dry Eyes and Asthenopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-0631
Record Dates: First submitted 2025-05-08; First posted 2025-05-28 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-05

CONDITIONS: Dry Eye Disease (DED); Asthenopia
MeSH Terms: conditions — Dry Eye Syndromes; Asthenopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- light condition (Sham Comparator): use smartphone under light condition for 45 minutes
  Interventions: Behavioral: using non-processing screens; Behavioral: using AR+CP screens
- dark condition (Experimental): use smartphone under dark condition for 45 minutes
  Interventions: Behavioral: using non-processing screens; Behavioral: using AR+CP screens

INTERVENTIONS:
Behavioral: using non-processing screens — ask subjects to use non-processing screens
Behavioral: using AR+CP screens — ask subjects to use AR+CP screens

SUMMARY:
This study aimed to evaluate the effect of anti-reflection (AR) and circularly polarized (CP) film on video display terminal (VDT) induced dry eye and asthenopia after limited time and close distance of visual tasks under light and dark environment, searching for new strategy for eye-protective electronic screen. The study was randomized, double-blind and controlled. Subjects were enrolled following the criteria: diopter of both eyes not exceeding -6.0D and anisometropia not exceeding 2.0D. and randomly divided into control, AR, AR+CP group in light or dark environment. Character searching, gaming and video tasks utilizing specific smartphones for totally 45 minutes were performed. Researchers measured the indexes of dry eye and asthenopia before and after tasks to evaluate impacts induced by VDT.

DETAILED DESCRIPTION:
The inclusion criteria required volunteers to have myopia diopter not exceeding -6.00D, hyperopia not exceeding +2.0D, astigmatism not exceeding -2.00D, anisometropia between both eyes not exceeding 2.00D. The key exclusion criteria were as follows: (1)strabismus and amblyopia; (2)used eye drops within 1 week; (3)had undergone eye surgery within 6 months; (4)worn contact lenses within the last 2 weeks; (5)had serious eye discomfort in the last 7 days; (6)Breastfeeding or pregnant women and patients with severe systemic diseases, psychosis or dementia.

Subjects who met the criteria were divided into five groups. 3 groups using non-processing smartphone screen, anti-reflection screen and anti-reflection plus circular polarization screen read in light environment and 2 groups using non-processing screen and anti-reflection plus circular polarization screen read in dark environment. Subjects did not know the characteristics of the smartphones they use. Subjects met the requirements were randomly grouped. The subjects did not use video terminals such as mobile phones within 30 minutes before the study began.

During the whole experiment, light-group subjects were in a room with normal indoor ceiling light, correlated colour temperature 3904K, desktop illuminance 388.7lux, screen brightness about 150nit, while dark-group in environment illuminance 0.02lux, screen brightness about 6nit. Light source stability (working surface illuminance fluctuation) greater than 99% during the whole experiment, desktop range uniformity greater than 80%. Desktop matte treatment without special reflection, indoor air conditioning control temperature: 22-25 degrees Celsius, humidity: 50-70%RH. Users placed it on a fixed mobile phone stand (the angle and height of the mobile phone stand can be adjusted to make sure all subjects could see reflection of the lamp on ceiling behind them from the smartphone black screen state). All subjects' eyes are 40cm away from the mobile phone screen, and they sit on a chair of appropriate height and fixed position. Two groups of subjects would complete the following three tasks in definite order: 1) Character searching task (5 minutes) : Subject read a meaningless text on the screen, found all the target characters in it, and told researchers about the statistics; 2) Game task: Subject played one of several pre-installed games requiring high concentration and eye tracking for 20 minutes; 3) Video task: Subject watched the video Animal World with the mobile phone for 20 minutes. During the study period, subjects should not do any behavior unrelated to watching the screen for a long time (more than 1 minute). We evaluated the subjects' basic ocular data: best corrected visual acuity(BCVA), spherical equivalent(SE), subjective questionnaires including Ocular Surface Disease Index(OSDI), Computer Vision Syndrome Scale 17 (CVSS17); dry eye comprehensive analysis before and after the experiment respectively: tear meniscus height(TMH), noninvasive tear break-up time(NIBUT), fluorescein tear break-up time(FBUT), corneal fluorescein staining(CFS), Schirmer I tear secretion test; asthenopia related examination: High-frequency component(HFC) and blink frequency.

ELIGIBILITY:
Inclusion Criteria:

* 1.have basic reading comprehension skills and to be older than 18 years old. 2.diopter of both eyes not exceeding -6.0D and anisometropia not exceeding 2.0D.

Exclusion Criteria:

* presbyopia or decreased regulation function, ocular inflammation and disease, worn contact lens within 1 month, history of eye surgery within 6 months, lactating or pregnant woman, have severe systemic diseases.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Flourescence tear break-up time | 2 months
  Drop a drop of physiological saline onto a sodium fluorescein test strip. Gently touch the middle of the conjunctiva of both lower eyelids of the examinee with the test strip respectively, and instruct the examinee to blink their eyes gently and look straight ahead. The examiner observed the tear film of the examinee with cobalt blue light under a slit lamp. The time of tear film rupture was the time from the examinee opening their eyes to the appearance of the first black spot on the tear film. Three TBUT tests were detected and recorded for each eye respectively, and the average and maximum values were taken.
HFC (high frequency component of accommodative fluctuation) | 2 months
  The SCR mode of the ACOMOREF K-MODEL computerized optometer was adopted. The subjects were asked to keep a close eye on the image. The image distance was gradually moved from infinity to 1m, 60cm, and 30cm, and remained at each of the four distances for 20 seconds. The equipment would analyze and record the high-frequency fluctuations of the subjects' ciliary muscles, known as HFC. After the test of the first eye, Take a 20-second break to test the second eye.
non-invasive tear break-up time | 2 months
  The Oculus ocular surface comprehensive analyzer was adopted. The examinees sat upright in front of the instrument and were asked to blink their eyes lightly and then look at the red marked object. The instrument automatically conducted ocular surface image analysis to obtain and record the first NIBUT and average NIBUT of the examinees

SECONDARY OUTCOMES:
tear meniscus height | 2 months
  The Oculus ocular surface comprehensive analyzer was used. The person being examined sat upright in front of the instrument and was asked to blink their eyes slightly and then look at the red marked object. The instrument automatically analyzed the ocular surface images to obtain the lacrimal river height data
corneal fluorescein staining | 2 months
  After character searching, gaming and video tasks utilizing specific smartphones for totally 45 minutes, CFS was measured.
computer vision symptom scale 17 | 2 months
  A subjective scale reflecting the symptoms of visual fatigue, including the occurrence frequency and intensity of 17 ocular and extraocular symptoms
Schirmer I test | 2 months
  The subjects were tested under non-anesthetic conditions. A 5mm×35mm filter paper was placed in the conjunctival sac of the inner 1/3 of the lower eyelid, with the remaining part hanging over the skin surface. The subjects were asked to gently close their eyes. After 5 minutes, the length of the filter paper soaked by tears was measured and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine (SAHZU), Hangzhou, Zhejiang, China